CLINICAL TRIAL: NCT05823467
Title: What is Optimal Post-operative Prophylactic Therapy in Irradiated Breasts Undergoing Repeat Oncologic Surgery to Reduce Early Wound Complications
Brief Title: What is Optimal Post-operative Prophylactic Therapy in Irradiated Breasts Undergoing Repeat Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0241
Record Dates: First submitted 2023-03-17; First posted 2023-04-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: radiation; breast conservation surgery; recurrent breast cancer; wound VAC; postoperative antibiotics; post operative wound complications; repeat breast surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: This study will randomize patients to three arms - patients will either be randomized to post operative antibiotic arm (1 week), post operative wound VAC arm (1 week), or no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post operative Antibiotic (Experimental): Patients in this arm will have a prescription for one week or post operative antibiotic ( 7-day course of TMP-SMX DS )
  Interventions: Drug: TMP-SMX DS
- Post operative Wound VAC (Experimental): Patient will have a 7-day application of ciNPT dressing post operatively.
  Interventions: Device: ciNPT dressing
- No Intervention (No Intervention): Patient will be treated as standard of care which is no intervention.

INTERVENTIONS:
Drug: TMP-SMX DS — Oral Antibiotic - used to treat post operative wound infections.
  Other Names: Trimethoprim / Sulfamethoxazole
  Arms: Post operative Antibiotic
Device: ciNPT dressing — Negative pressure wound VAC placed on incision post operatively.
  Other Names: PICO dressing
  Arms: Post operative Wound VAC

SUMMARY:
This study will look at whether females who have previously had breast surgery and radiation and are undergoing repeat breast surgery require any post operative interventions. The reason the investigators are conducting this study is because females who have undergone breast radiation are at higher risk of wound complications following breast surgery. The investigators will randomize recruited female participants into three arms, one which is post operative antibiotics for one week, one which is a wound VAC, and one which is no intervention. The investigators goal is to identify whether these patients will require any postoperative interventions.

DETAILED DESCRIPTION:
Background:

The 10-year local recurrence rate for breast cancer following breast conserving surgery (BCS) and radiation therapy (RT) is estimated around 19% for which the standard of care is completion mastectomy. This represents a growing population of patients with prior irradiation undergoing repeat oncologic surgery. Patients undergoing surgery after RT have been shown to be at higher risk for wound complications such as surgical site infection (SSI), dehiscence, and skin necrosis. The average rate of SSI following major breast surgery is estimated at 5%, whereas it has been reported over 30% in irradiated patients. However, the data remains sparse dedicated to mitigating early wound complications in this patient population with guidelines or recommendations that exist for prophylactic measures.

A retrospectively review analyzed SSI rate in patients undergoing mastectomy without reconstruction and found a statistically significant reduction in SSI rate with post-operative antibiotics in the subset of patients with previous RT (30.8% to 3.6%). In another study of a prospectively followed cohort of high-risk patients undergoing breast cancer surgery, a subset of whom had previous RT, these patients were found to have a significant reduction from 45% to 4% for all wound complications (no reported SSI) with closed incision negative pressure wound therapy (ciNPT) and post-operative antibiotics. Therefore, the investigators hypothesize that patients with prior BCS and RT undergoing repeat oncologic breast surgery would benefit from post-operative prophylactic therapy to reduce early wound complications. Retrospective analyses and prospective cohort studies have demonstrated potential benefit; however, a high quality RCT is warranted to analyze our research question.

Study Design:

The investigator's primary objective will be to evaluate the effect of a 7-day course of TMP-SMX DS and 7-day application of ciNPT dressing (PICO) on the rate of early wound complications in this patient population. This study will be designed as an unblinded block randomized controlled trial with three arms: 1) standard of care 2) post-operative antibiotics 3) ciNPT. Participants will be recruited by surgeons at the Meadowlark and Sturgeon surgical clinics. Data will be collected via paper forms or Connect Care at 1-2 week and 4-6 week post-operative visits. The primary outcome measure will be wound complications (SSI, dehiscence, skin necrosis). Secondary outcomes will include adverse effects of antibiotics or ciNPT therapy, and other post-operative complications (extended antibiotic therapy, re-operation, admission to hospital).

Impact:

The investigators hope the results of this trial will demonstrate benefit of prophylactic antibiotics and/or ciNPT to decrease wound complications in this patient population. This will have the potential to create recommendations for a post-operative prophylactic regimen to inform future guidelines and practice in oncologic breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* > 18 years of age
* Previous breast surgery and ipsilateral breast irradiation
* Requiring repeat breast surgery

Exclusion Criteria:

* Male
* <18 years of age,
* Currently on antibiotic therapy for other indications
* Known hypersensitivity to trimethoprim or sulfonamides,
* History of drug-induced immune thrombocytopenia with use of trimethoprim and/or sulfonamides
* Documented megaloblastic anemia due to folate deficiency
* Currently pregnant or breastfeeding, and
* Marked hepatic damage
* Severe renal insufficiency
* Severe sensitivity or allergy to silicone adhesive

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with Breast Cancer - male breast cancer will present a confounding variable
Enrollment: 105 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound Complication | Post operative day 14 during follow up visit
  Assessment of rate of Wound complication with each intervention arm, immediately after intervention

SECONDARY OUTCOMES:
Adverse effects from intervention arm | post procedure from post operative day 1 - post operative day 30
  Will assess for any adverse reaction from each intervention as well as repeat hospital visit within 30 days (after the procedure and intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Rajaee, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Meadowlark Health Centre, Edmonton, Alberta
  - St Thomas Surgical Clinic, St. Albert, Alberta

REFERENCES:
- [Background] Edwards BL, Stukenborg GJ, Brenin DR, Schroen AT. Use of prophylactic postoperative antibiotics during surgical drain presence following mastectomy. Ann Surg Oncol. 2014 Oct;21(10):3249-55. doi: 10.1245/s10434-014-3960-7. Epub 2014 Aug 20. PMID 25138078
- [Background] Ferrando PM, Ala A, Bussone R, Bergamasco L, Actis Perinetti F, Malan F. Closed Incision Negative Pressure Therapy in Oncological Breast Surgery: Comparison with Standard Care Dressings. Plast Reconstr Surg Glob Open. 2018 Jun 15;6(6):e1732. doi: 10.1097/GOX.0000000000001732. eCollection 2018 Jun. PMID 30276035
- [Background] Olsen MA, Nickel KB, Margenthaler JA, Wallace AE, Mines D, Miller JP, Fraser VJ, Warren DK. Increased Risk of Surgical Site Infection Among Breast-Conserving Surgery Re-excisions. Ann Surg Oncol. 2015;22(6):2003-9. doi: 10.1245/s10434-014-4200-x. Epub 2014 Oct 31. PMID 25358666
- [Background] Ruvalcaba-Limon E, Robles-Vidal C, Poitevin-Chacon A, Chavez-Macgregor M, Gamboa-Vignolle C, Vilar-Compte D. Complications after breast cancer surgery in patients treated with concomitant preoperative chemoradiation: A case-control analysis. Breast Cancer Res Treat. 2006 Jan;95(2):147-52. doi: 10.1007/s10549-005-9058-y. Epub 2005 Dec 1. PMID 16319989